CLINICAL TRIAL: NCT00204971
Title: Randomized, Placebo-controlled Clinical Trial of Enteral Glutamine Supplementation in Neurologically-injured Patients
Brief Title: Enteral Glutamine in Neurologically-injured Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 2002-0409
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Neurologic Injury; Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Nutritional supplement
  Interventions: Dietary Supplement: Enteral glutamine powder
- 2 (Placebo Comparator): placebo
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: Enteral glutamine powder — nutritional supplement
  Arms: 1
Other: placebo — placebo control
  Arms: 2

SUMMARY:
Nutrition is an important part of the recovery process after having a head injury so that subjects can gain strength and fight off infection. Liquid nutrition formulas are often given to patients through a tube that has been placed into the intestines for feeding when they are unable to eat on their own. Some reports suggest that nutrition with extra amounts of the amino acid called glutamine may decrease infections and hospital stay in severely injured patients.The purpose of this study is to evaluate if giving extra amounts of an amino acid called glutamine with liquid nutrition formulas will decrease the risk of infection and length of stay in the intensive care unit after having a head injury.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Nonpregnant females
* Aged 18-75 years old
* Glasgow Coma Scores of 3-12
* Injury Severity Scores greater than or equal to 20
* Requiring enteral nutrition for a minimum of 5 days

Exclusion Criteria:

* Documented hepatic dysfunction
* Acute renal failure (creatinine clearance < 15 mL/min)
* Gastrointestinal malabsorptive disorder
* Infection at time of admission

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2003-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Nosocomial infections | throughout study

SECONDARY OUTCOMES:
Multiple organ dysfunction syndrome | throughout the study
Nutritional outcome parameters | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Gordon S Sacks, PharmD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States